CLINICAL TRIAL: NCT02957851
Title: Equimolar Mixture of Oxygen and Nitrous Oxide (EMONO) for the Treatment of Peripheral Neuropathic Pain: A Randomises, International, Multicentre, Placebo-Controlled, Phenotype-stratified Phase IIa Study
Brief Title: EMONO for the Treatment of Peripheral Neuropathic Pain
Acronym: ProtoTOP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Air Liquide Santé International (Industry)
Collaborators: AMS Advanced Medical Services GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALMED-15-C2-054
Record Dates: First submitted 2016-10-20; First posted 2016-11-08 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Neuralgia
MeSH Terms: conditions — Neuralgia | interventions — Air; Oxygen; Nitrogen; Nitrous Oxide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxygen/Nitrogen (22%/78%) (Placebo Comparator): Medical Air
  Interventions: Drug: Medical Air
- Nitrous Oxide/Oxygen (50%/50%) (Active Comparator): EMONO
  Interventions: Drug: EMONO

INTERVENTIONS:
Drug: Medical Air
  Other Names: Oxygen/Nitrogen
  Arms: Oxygen/Nitrogen (22%/78%)
Drug: EMONO
  Other Names: Nitrous Oxide/Oxygen
  Arms: Nitrous Oxide/Oxygen (50%/50%)

SUMMARY:
To assess the effect of 3 consecutive days of one-hour administration of Nitrous Oxide/Oxygen 50%/50% (EMONO) versus placebo as Oxygen/Nitrogen 22%/78% (synthetic medical air), in add-on therapy to chronic analgesic treatments, on average pain intensity in patients with chronic peripheral neuropathic pain. A total of 250 randomised patients to be included in all the participating centres, i.e., 125 randomised patients in each of the 2 study groups treatments

ELIGIBILITY:
Inclusion Criteria:

* Patients with a mean pain intensity from 4 to 9 as assessed daily with a Numerating Rating Scale during the 7 day period preceding inclusion in spite of administration of usual pain treatments.
* Neuropathic pain lasting for more than 3 months but less than 10 years
* Definite or probable peripheral neuropathy

Exclusion Criteria:

* legal incapacity
* patient with another concomitant chronic pain
* ongoing major depression
* Chemotherapy-induced peripheral neuropathic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2016-11; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 7 days after the last administration of treatment
  Numeric Rating Scale (NRS)

SECONDARY OUTCOMES:
Pain intensity | 28 days after the last administration of treatment
  Numeric Rating Scale (NRS)
Pain characteristic | 28 days after the last administration of treatment
  Neuropathic Pain Symptom Inventory (NPSI)
Quality of life questionnaire | 28 days after the last administration of treatment
  Medical Outcome Study Short Form (SF-12)
Number of patients with adverse events | through study duration, up to 31 days

CONTACTS AND LOCATIONS:
Overall Officials: Didier Bouhassira, MD, Study Chair — Hospital Ambroise Paré Paris
Locations (22):
- France (20):
  - CHU de Grenoble, Grenoble, La Tronche
  - Centre Hospitalier de Bayeux, Bayeux
  - Centre Hospitalier Regional Universitaire - Hôpital Jean-Minjoz, Besançon
  - Hôpital Pellegrin, Bordeaux
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - Hopital Neurologique Weirthermer, Bron
  - Centre Hospitalier Universitaire Gabriel Montpied, Clermont-Ferrand
  - Clinique du Bourget, Le Bourget
  - Centre Hospitalier Universitaire Dupuytren, Limoges
  - CHU la Timone, Marseille
  - Centre Hospitalier Régional de Metz-Thionville, Metz-Thionville
  - Hôpital Saint Eloi, Montpellier
  - Clinique Brétéché, Nantes
  - Hôpital Nord Laennec, Nantes
  - Nouvelles Cliniques Nantaises, Nantes
  - Hôpital Universitaire Caremeau, Nîmes
  - Hôpital Lariboisière, Paris
  - Hôpital Cochin, Paris
  - Centre hospitalier Universitaire de Rouen, Rouen
  - Clinique IRIS Saint-Priest, Saint-Priest
- Germany (2):
  - Neurologische Klinik Universitätsklinikum, Würzburg, Josef-Schneider-Str. 11
  - Neurologische Klinik Klinikum rechts der Isar, München

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bouhassira D, Perrot S, Attal N, Ramirez-Gil JF, Delval C, Schaller M, Bessiere B, Houeto P, Sommer C. Combination of inhaled nitrous oxide and oral opioids induces long-lasting analgesic effects in patients with neuropathic pain: ProtoTOP study post hoc exploratory analyses. Pain. 2022 Sep 1;163(9):e1021-e1029. doi: 10.1097/j.pain.0000000000002570. Epub 2021 Dec 20. PMID 35050957
- [Derived] Bouhassira D, Perrot S, Riant T, Martine-Fabre G, Pickering G, Maindet C, Attal N, Ranque Garnier S, Nguyen JP, Kuhn E, Viel E, Kieffert P, Tolle T, Delorme C, Deleens R, Ginies P, Corand-Dousset V, Dal-Col C, Serrie A, Chevrillon E, Gov C, Ramirez-Gil JF, Delval C, Schaller M, Bessiere B, Houeto P, Sommer C; ProtoTOP group. Safety and efficacy of an equimolar mixture of oxygen and nitrous oxide: a randomized controlled trial in patients with peripheral neuropathic pain. Pain. 2021 Apr 1;162(4):1104-1115. doi: 10.1097/j.pain.0000000000002109. PMID 33044394